CLINICAL TRIAL: NCT06262321
Title: Phase II Trial of Thoracic Radiotherapy for Patients With Metastatic (Stage IV) Non-Small Cell Lung Cancer at High Risk of Symptomatic Progression Within the Thorax
Brief Title: Thoracic Radiotherapy for Patients With Metastatic (Stage IV) Non-Small Cell Lung Cancer at High Risk of Symptomatic Progression Within the Thorax
Acronym: DRO2301
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Michael Milano, MD,PhD, Michael Milano, Assistant Professor of Radiation Oncology at the University of Rochester School of Medicine and Dentistry, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: URLUN23099
Record Dates: First submitted 2024-02-07; First posted 2024-02-16 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Stage 4 NSCLC; Radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prophylactic Palliative Radiotherapy (Experimental): Prophylactic Palliative Radiotherapy
  Interventions: Radiation: Prophylactic Palliative Radiotherapy

INTERVENTIONS:
Radiation: Prophylactic Palliative Radiotherapy — Prophylactic Palliative Radiotherapy

SUMMARY:
Patients with metastatic non small cell lung cancer with high risk location or size are treated with prophylactic radiation therapy in conjunction with standard of care systemic therapy.

DETAILED DESCRIPTION:
This will be a single-cohort Phase II single center, prospective trial. Patients with stage IV NSCLC are eligible. Patients may receive standard of care systemic therapy (chemotherapy and/or immunotherapy). Radiotherapy will be directed at high-risk disease (primary cancer, nodal metastases, and metastases) in the thorax. Treatment of other sites of extrathoracic metastases would be allowed as per standard of care. Standard chest radiation dosing and normal tissue exposures (based on published or ongoing studies) will be applied. There is no plan to escalate the chest radiation dose (i.e., no Phase I component) as palliative regimens for NSCLC have been routinely used for many decades.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of Non-Small Cell Lung Cancer (NSCLC) without targetable/oncogene driven mutations (i.e., EGFR mutations, ALK-rearrangement, ROS1 rearrangement).
* T1-4(or Tx)N0-3M1a-c, Stage IV disease (using the 8th edition of the AJCC staging manual) or metastatic recurrence of primary Stage I-III NSCLC that had been treated with curative intent therapy, without prior thoracic radiotherapy.
* Thoracic lung and/or nodal lesion(s) amenable to palliative chest radiotherapy.
* All subjects are required to have one or more of the following high-risk features: a) a non-central primary lung lesion ≥5 cm in size (at least T3 by criteria); b) bulky (≥2 cm) parenchymal lung lesions and/or nodal lesions abutting (within 1 cm) any of the following: Proximal bronchial tree, Esophagus, Vertebra, Heart, brachial plexus or subclavian vessels (if brachial plexus not well visualized), Superior vena cava
* Prior systemic therapy is allowed. Subjects must be enrolled within 6 months of first cycle of systemic therapy for Stage IV disease.
* Systemic therapy following the thoracic radiotherapy (on protocol) is allowed.
* Prior palliative surgical treatment (including airway debridement) is allowed.
* Concurrent chemotherapy (chemotherapy delivered from ≤2 days of before through ≤2 days after radiotherapy) is NOT allowed.
* Concurrent immunotherapy therapy is allowed.
* Subjects may undergo (or may have undergone) standard extrathoracic radiotherapy off protocol, including (but not limited to): Palliation of symptomatic bone metastases, prophylactic palliation of high-risk bone metastases, cranial radiosurgery (with controlled intracranial metastases if performed prior to enrollment), Ablative or non-ablative definitive radiotherapy for oligometastases.
* Subjects may undergo concurrent palliative thoracic radiotherapy (per study) and palliative radiotherapy for thoracic bone metastases (i.e., painful spine or rib metastases). It is anticipated that the study will be open at multiple sites within the Wilmot Cancer Institute network. Among these sites, subjects may be consulted and consented at any site, simulated and planned at any site, and treated at any site (even if different from the site(s) at which the subject was consulted and simulated).

Exclusion Criteria:

* Prior radiation therapy to the thoracic region.
* Active systemic lupus or Sjogren's disease.
* NSCLC (primary, nodal sites or metastases) causing severe symptoms requiring thoracic palliative radiotherapy for indications other than bone pain. These symptoms include superior vena cava syndrome, active and large volume (>100 ml per day) hemoptysis, airway obstruction (stridor, post-obstructive pneumonia, progressive dyspnea not attributed to other causes), compression of the spinal cord or spinal nerve roots, vertebral compression fracture, brachial plexopathy (from compression).
* Baseline ECOG performance status of 3-4. For the purposes of eligibility, Karnofsky Performance Score (KPS) will be converted to ECOG/Zubrod performance score, per ECOG guidelines.
* Brain metastases not amenable to immunotherapy alone, resection or stereotactic radiosurgery (i.e., brain metastases requiring whole brain radiotherapy).
* Malignant pleural effusion attributable to grossly apparent pleural disease. Subjects with malignant pleural effusion amenable to therapeutic thoracenteses and without radiographic evidence of pleural disease (i.e., studding or masses) are potentially eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from symptomatic progression of irradiated thoracic target(s) | 6 month, 1 year, and 2 years
  Kaplan-Meier freedom from symptomatic progression of irradiated thoracic target(s) at 6 months, 1 year, and 2 years.

SECONDARY OUTCOMES:
OS (Kaplan-Meier) (Kaplan-Meier) | 6 month, 1 year, and 2 years
  Kaplan Meier Overall Survival
Freedom from local recurrence of irradiated thoracic target lesion(s) | 6 month, 1 year, and 2 years
  Freedom from local recurrence of irradiated thoracic target lesion(s)
PFS (freedom from local and distant progression; Kaplan-Meier) | 6 month, 1 year, and 2 years
  Progression (local or distant) free survival Outcome
Duration of time that patient is maintenance | 6 month, 1 year, and 2 years
  Duration of time that patient remains on maintenance systemic therapy

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided